CLINICAL TRIAL: NCT05238350
Title: The Effect of Acupressure on Pain, Functional Status and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: The Effect of Acupressure in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Pınar TEKİNSOY KARTIN (Unknown); Rabiye ÇIRPAN (Unknown)
Responsible Party: Principal Investigator, Tuğba AYDEMİR, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NevsehirU
Record Dates: First submitted 2021-12-21; First posted 2022-02-14 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Pain; Nursing; Acupressure.
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: The study was conducted as an experimental study with a pre-posttest and a control group.
Who Masked: Participant

ARMS (2):
- Acupressure (intervention group) (Experimental): The intervention group was performed with 45 patients. Acupressure was performed two days a week for four weeks with a total of eight sessions on the ST34, ST35, ST36, SP9, SP10, GB34 acupuncture points following an acupressure practice guide prepared by the researcher.
  Interventions: Procedure: Acupressure
- Control group (No Intervention): Thecontrol group was performed with 45 patients. Any application was not performed for the control group.

INTERVENTIONS:
Procedure: Acupressure — Acupressure was performed two days a week for four weeks with a total of eight sessions on the ST34, ST35, ST36, SP9, SP10, GB34 acupuncture points following an acupressure practice guide prepared by the researcher.
  Other Names: Control
  Arms: Acupressure (intervention group)

SUMMARY:
Abstract Pain is the most common symptom of osteoarthritis and affects people's functional status with quality of life. This study was conducted to determine the effect of acupressure on pain, functional status, and quality of life in patients living with knee osteoarthritis. Acupressure application and follow-ups were performed by the researcher in the patient's home environment. The study was performed with 90 patients, 45 in the intervention group and 45 in the control group. Acupressure was performed two days a week for four weeks with a total of eight sessions on the ST34, ST35, ST36, SP9, SP10, GB34 acupuncture points following an acupressure practice guide prepared by the researcher. It was determined that while the Visual Analog Scale (VAS), the Western Ontario and McMaster University Osteoarthritis Index (WOMAC) scores of the intervention group were higher than those of the control group before application, they had decreased after application. It was found that all subscale mean scores of the Short-Form Health Survey (SF-36) quality of life questionnaire increased after application in the intervention group. It was concluded that acupressure has decreased pain severity and increased the functional status and quality of life of patients with knee osteoarthritis.

Keywords: Osteoarthritis, pain, nursing, acupressure.

DETAILED DESCRIPTION:
Abstract Background: Pain is the most common symptom of osteoarthritis and affects people's functional status with quality of life.

Objective: This study was conducted to determine the effect of acupressure on pain, functional status, and quality of life in patients living with knee osteoarthritis.

Methods/Design: The study was conducted as an experimental study with a pre-posttest and a control group.

Settings: The study was conducted on patients diagnosed with knee osteoarthritis and attended the Physical Therapy and Rehabilitation Polyclinics of Nevşehir government hospital in the Central Anatolia Region of Turkey. Acupressure application and follow-ups were performed by the researcher in the patient's home environment.

Participants: The study was performed with 90 patients, 45 in the intervention group and 45 in the control group.

Intervention: Acupressure was performed two days a week for four weeks with a total of eight sessions on the ST34, ST35, ST36, SP9, SP10, GB34 acupuncture points following an acupressure practice guide prepared by the researcher.

Measurement of efficacy: Data was collected before and after acupressure application by using a Visual Analogue Scale (VAS), the 36-Item Short-Form Health Survey (SF-36), and the Western Ontario and McMaster University Osteoarthritis Index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

* 38 years old and over
* Diagnosed by a doctor with knee OA according to American College of Rheumatology (ACR) criteria
* had three points and over on the VAS pain scale,
* had no communication problems
* did not have any significant knee trauma within the last six months or an intra-articular steroid injection
* did not have any infection in the lower extremities or wounds, surgery or physiotherapy within the last six months
* those who accepted to participate to the study.

Exclusion Criteria:

* the patient is not willing to go on the study in any stage of the study and case of any adverse effect of acupressure.

Min Age: 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-03-07 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2015-11-11 (Actual)

PRIMARY OUTCOMES:
Pain level in visual analogue scale (VAS) | baseline, change from baseline at 4th week;
  Pain severity scores were determined by measuring values that were chosen on VAS by patients. The numerical scale ranges from 0 "No pain", to 10 "Worst pain imaginable", and a numerical value is given to every 1 cm range to measure pain severity.

SECONDARY OUTCOMES:
The Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Osteoarthritis Index | baseline, change from baseline at 4th week;
  Their functional status levels were evaluated by using WOMAC Osteoarthritis Index.Every question is scored between 0 and 4 points evaluated with a five-way Likert-type scale. High scores from the index show increased pain and stiffness and dysfunction in physical function.
36-Item Short-Form Health Survey (SF-36) | baseline, change from baseline at 4th week;
  Their changes in quality of life levels were evaluated by using SF-36 scale.The scale gives separate scores for every sub-scale, which varies between 0 and 100 points. High scores on the subscales show good health status, while low scores show a deterioration in health

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba AYDEMİR, RN, MSc, Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Ni̇ğde, Turkey (Türkiye)

REFERENCES:
- [Derived] Aydemir T, Cirpan R, Tekinsoy Kartin P. Impact of Acupressure on Pain, Functional Status, and Quality of Life in Individuals With Knee Osteoarthritis. J Manipulative Physiol Ther. 2025 Jan-Jun;48(1-5):204-213. doi: 10.1016/j.jmpt.2025.09.001. Epub 2025 Oct 7. PMID 41055613